CLINICAL TRIAL: NCT03986294
Title: A Randomized Phase II Study of Second Line Treatment With Liposomal Irinotecan and S1 Versus Liposomal Irinotecan and 5-fluorouracil in Patients With Metastatic Pancreatic Cancer Who Failed on First Line Gemcitabine-based Chemotherapy
Brief Title: Second Line Treatment With Nal-IRI and S1 in Pancreatic Cancer
Acronym: NAPAN
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: UMC Utrecht (Other); Isala (Other); Maastricht University Medical Center (Other); Vall de Hebron, Barcelona, Spain (Unknown); University Hospital Verona, Italy (Unknown); Odense University Hospital (Other); Medical University of Vienna (Other)
Responsible Party: Principal Investigator, J.W. Wilmink, Principle investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL64126.018.17
Record Dates: First submitted 2019-02-11; First posted 2019-06-14 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: Liposomal irinotecan; S1; Pancreatic cancer; Second line
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — S 1 (combination); irinotecan sucrosofate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- S1 and liposomal irinotecan (Experimental): S-1 will be given for 14 consecutive days, twice daily, followed by 2 weeks rest. Nal-IRI will be administered as an iv infusion on day 1 and 15. Treatment will be repeated every 4 wks.
  Interventions: Drug: S1 + Nal-IRI; Drug: Nal-IRI+Leucovorin+5-FU
- Liposomal irinotecan, Leucovorin and 5-fluoracil (Experimental): Nal-IRI 80 mg/m2 administered first, followed by LV 400 mg/m2, followed by 5-FU 2400 mg/m2 as an IV infusion over 46-hrs on days 1-3. Each cycle consists of 14 days. Treatment will be repeated every 2 wks.
  Interventions: Drug: Nal-IRI+Leucovorin+5-FU

INTERVENTIONS:
Drug: S1 + Nal-IRI — S-1 will be given for 14 consecutive days, twice daily, followed by 2 weeks rest. Nal-IRI will be administered as an intravenous infusion on day 1 and 15. Courses of treatment will be repeated every 4 weeks.
  Arms: S1 and liposomal irinotecan
Drug: Nal-IRI+Leucovorin+5-FU — Nal-IRI 80 mg/m2 will be administered first, followed by LV 400 mg/m2, followed by 5-FU 2400 mg/m2 as an IV infusion over 46-hours on days 1-3. Each cycle consists of 14 days. Courses of treatment will be repeated every 2 weeks.

SUMMARY:
To determine the optimal second line treatment strategy in patients with metastatic pancreatic cancer who underwent a therapy with gemcitabine.

DETAILED DESCRIPTION:
The 5-year survival of patients with pancreatic cancer is less than 5%. Despite improvements over the past years with the introduction of FOLFIRINOX (5-fluorouracil, irinotecan, oxaliplatin and leucovorin) and gemcitabine and nab-paclitaxel, the vast majority will have disease recurrence or progression within 6 months. Single-arm phase II studies have been conducted after gemcitabine-based therapy. Randomized clinical trial data are limited in this setting, but the conclusion up to recently was that there is no superior chemotherapeutic regimen after gemcitabine failure. However, the NAPOLI trial altered the treatment landscape. In this trial, patients with metastatic pancreatic cancer that progressed after treatment with gemcitabine-based chemotherapy received liposomal irinotecan (nal-IRI) either as single agent or in combination with 5-fluorouracil/ leucovorin (5-FU/LV), or 5-FU/LV alone. Patients treated with the combination of nal-IRI plus 5-FU/LV experienced a median survival of 6.1 months versus 4.2 months for the 5-FU/LV group.

Recently, two studies on the clinical use of S-1 for pancreatic cancer have been reported from Japan. In the first study, S-1 demonstrated non-inferiority to gemcitabine in overall survival (OS) for advanced pancreatic cancer. In the second study, S-1 showed superiority to adjuvant chemotherapy with gemcitabine in OS. In addition to gemcitabine, S-1 is now regarded as the key drug in the management of pancreatic cancer in Japan. Phase II studies of S-1 in patients with gemcitabine-resistant pancreatic cancer have demonstrated moderate activity with acceptable toxicity. Although there has been no confirmed evidence based on phase III trials, S-1 would be a feasible treatment option in this patient population.

Objective:

To determine the optimal second line treatment strategy in patients with metastatic pancreatic cancer, whereby the hypothesis is, based on studies conducted in the Asian population, that the combination of S-1 and nal-IRI will be superior compared to 5-FU/ LV and nal-IRI, in terms of progression free survival. Therefore, patients will be randomized, after the optimal dose of S-1 and nal-IRI has been determined in the run in phase, between S-1 in combination with nal-IRI and 5-FU/LV in combination with nal-IRI during the phase II part of the study.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy all of the following inclusion criteria to be enrolled in the study.

1. Able to understand and provide written informed consent
2. ≥ 18 years of age
3. Histologically or cytologically confirmed adenocarcinoma of pancreas
4. Documented metastatic disease, according to RECIST 1.1.
5. Previously treated with gemcitabine or gemcitabine containing therapy, or progression within 6 months of adjuvant gemcitabine based treatment
6. Adequate hepatic, renal and hematological function

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

1. Serum total bilirubin ≥1.5 x ULN (biliary drainage is allowed for biliary obstruction)
2. Severe renal impairment (CLcr ≤ 30 ml/min)
3. Inadequate bone marrow reserves as evidenced by:

   1. ANC ≤ 1,5 x 10 9 /L; or
   2. Platelet count ≤ 100 x 10 9 /L;
4. WHO/PS 0-1
5. Any clinically significant disorder impacting the risk-benefit balance negatively per physician's judgment
6. Any clinically significant gastrointestinal disorder, including hepatic disorders, bleeding, inflammation, occlusion, or diarrhea > grade 1
7. Severe arterial thromboembolic events (myocardial infarction, unstable angina pectoris, stroke) in last 6 months
8. NYHA Class III or IV congestive heart failure, ventricular arrhythmias or uncontrolled blood pressure. Or known abnormal ECG with clinically significant abnormal findings
9. Active infection or an unexplained fever >38.5°C (excluding tumor fever), which in the physician's opinion might compromise the patient's health
10. Current use or any use in last two weeks of strong CYP3A-enzyme inducers/inhibitors and/or strong UGT1A inhibitors
11. Known hypersensitivity to any of the components of liposomal irinotecan (Nal-IRI) other liposomal irinotecan formulations, irinotecan, fluoropyrimidines, or leucovorin.
12. Hypersensitivity to any of the active substances (tegafur, gimeracil, and oteracil)
13. Previous treatment with fluoropyrimidine therapy
14. Known dihydropyrimidine dehydrogenase (DPD) deficiency
15. Breast feeding, known pregnancy, positive serum pregnancy test or unwillingness to use a reliable method of birth control, during therapy and for 3 months following the last dose of liposomal irinotecan (Nal-IRI).

Treatment within 4 weeks with DPD inhibitors, including sorivudine or its chemically related analogues such as brivudine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
DLT of Nal-IRI with S1 | 36 months
  Dose limiting toxicity (DLT) of nal-IRI when co-administered with fixed dose S1 in patients with metastatic pancreatic cancer
MTD of Nal-IRI with S1 | 36 months
  Maximum tolerated dose (MTD) of nal-IRI when co-administered with fixed dose S1 in patients with metastatic pancreatic cancer
Progression free survival of NaI-IRI with S1 | 36 months
  Determination of the efficacy between the treatment arms in terms of progression free survival.

SECONDARY OUTCOMES:
Overall survival | 36 months
  To determine the overall survival (OS) benefit of nal-IRI combined with S-1, compared with nal-IRI combined with 5-FU/LV, in subjects pre-treated with gemcitabine based chemotherapy for metastatic pancreatic ductal adenocarcinoma.
Response rate according to RECIST 1.1 | 36 months
  To determine the response rate according to RECIST 1.1 of nal-IRI combined with S-1, compared with nal-IRI combined with 5-FU/LV, in subjects pre-treated with gemcitabine based chemotherapy for metastatic pancreatic ductal adenocarcinoma.
Adverse events according NCI CTC version 4.0 | 36 months
  To determine the adverse events according to NCI CTC version 4.0 of nal-IRI combined with S-1, compared with nal-IRI combined with 5-FU/LV, in subjects pre-treated with gemcitabine based chemotherapy for metastatic pancreatic ductal adenocarcinoma.
Quality of life QoL (QLQ-C30) | 36 months
  To determine Quality of life (QoL) benefit of nal-IRI combined with S-1, compared with nal-IRI combined with 5-FU/LV, in subjects pre-treated with gemcitabine based chemotherapy for metastatic pancreatic ductal adenocarcinoma using a questionnaire QLQ-C30.Scale ranges 1-4, 1 is very good, 4 is very bad. Higher values represent a worse outcome.

OTHER OUTCOMES:
stromal markers | 36 months
  To assess expression of relative abundance of stroma in metastatic tumor tissue and stromal markers, including ADAM12 in metastatic tumor tissue and blood as predictor of response to treatment and survival.
Imaging (MRI) | 36 months
  To explore, by imaging the number of participants with the effects of the treatment combination on tumor vascularity, and stromal density.
ctDNA | 36 months
  To explore the number of participants with changes in ctDNA.

CONTACTS AND LOCATIONS:
Overall Officials: J W Wilmink, MD, PhD, Principal Investigator — Ademic Medical Center Amsterdam
Locations (1):
- Academic Medical Center, Medical Oncology, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No